CLINICAL TRIAL: NCT03615547
Title: Interest of Clomiphene Citrate (CC) Associated With a Second Testicular Sperm Extraction (TESE) in Patients With Non-obstructive Azoospermia (NOA) After Failure of a First TESE, on the Quantity of Sperm Cells Available for Intracytoplasmic Sperm Injection (ICSI). Randomized Double Blind Trial Versus Placebo.
Brief Title: Interest of Clomiphene Citrate in Patients With Non-obstructive Azoospermia on the Quantity of Sperm Cells
Acronym: CLOMINOA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL18_0033
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Azoospermia, Nonobstructive
Keywords: azoospermia; clominophene
MeSH Terms: conditions — Azoospermia, Nonobstructive; Azoospermia | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clomifene citrate group (Experimental): a daily dose of 50mg of Clomifene Citrate per os during 9 months
  Interventions: Drug: Clomifene Citrate
- Placebo group (Experimental): a daily dose of 50mg per os of placebo (lactose monohydrate) during 9 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clomifene Citrate — After randomization, the andrologist will give a prescription with the first three months of treatment (Clomifene Citrate or placebo) to be collected to the local hospital pharmacy. The andrologist will be blind of the treatment arm.
  Treatment unit and their shipment to local pharmacy will be provided and organized by the East group pharmacy of the Hospices Civils of Lyon which is the coordination pharmacy for this study. Prescription and delivery will be renewed for three months at the 3 month and 6 months visit.
  The experimental treatment consists in a daily dose of 50mg of Clomifene Citrate per os during 9 months followed by a second TESE if no spermatozoid has been obtained from semen. The dose level was set according to Chua et al 2013 (cf 1.2.2). One capsule containing 50 mg of CC will be orally administered in the morning every day.
  Arms: Clomifene citrate group
Other: Placebo — The placebo treatment consists in a daily dose of 50mg of lactose monohydrate per os during 9 months followed by a second TESE if no spermatozoid has been obtained from semen. The capsule containing the placebo will have the exact same size, weight, color, taste and will be delivered in the exact same condition as the experimental treatment capsule.
  Arms: Placebo group

SUMMARY:
In the absence of sperm in the semen (azoospermia), there is no chance of natural paternity. It is found in about 1% of men and is either due to an obstruction of the seminal tracks (obstructive azoospermia (OA)) in 1/3 of the cases, or a spermatogenic failure (non-obstructive azoospermia (NOA)) in 2/3 of the cases. To date, no medical treatment had proved its efficiency to induce spermatogenesis in case of NOA.

The development of Intracytoplasmic sperm injection (ICSI) in 1992 allowed to obtain pregnancies from a small number of spermatozoa. The next year, testicular sperms were extracted from testicular tissue obtained surgically in cases of OA , allowing paternity for azoospermic men. In case of NOA, TESE allowed to obtain few sperms in an unexpected number of cases. It was shown that spermatogenesis remains active in rare portions of seminiferous tubules, a phenomenon called focal spermatogenesis, which allows to extract testicular sperms with an average SRR of 50%, and to obtain pregnancy by ICSI. Thus, TESE-ICSI revolutionized the prognosis of NOA, however, half of the cases of NOA had no sperm extracted and remained sterile . Since sperm donation and adoption are unacceptable for several of these couples, there is a real demand for additional treatment.

Two ways to improve chances of paternity in case of NOA are currently discussed:

1. Proceed to a second attempt of TESE. Since the first attempt could have missed a focus of active spermatogenesis, the chance for a positive second TESE is not null even. Reviewing the few articles published on this issue , the SRR for the second attempt, after a first negative attempt averaged 25%.
2. Based upon the decrease of testosterone production within the testis in case of NOA and the potential increased of the focal spermatogenesis by gonadotropins, few reports of hormonal therapy in case of NOA have been published and suggested a positive effect of hormonal therapy.

This prompted us to develop this clinical trial to investigate the effect of Clomiphene Citrate versus placebo on the results of a second TESE in NOA.

Results of hormonal therapy in case of NOA were heterogeneous and of poor methodological quality, none was randomized versus placebo: Anti-aromatases or Gonadotropins administered before the first TESE or the second TESE gave positive results. Hussein at al in 2013, suggested a positive effect of Clomiphene citrate (CC), administrated before the first TESE (57% of the CC treated group versus 33.6% in not treated group) but with drop out of patient positive to sperm analysis. However, in these positive studies, sample sizes were small or selected patients on hormonal status or histology criteria suggesting subgroup of favourable NOA. Thus, there is no strong evaluation of the interest of hormonal treatment in NOA, after a negative first TESE.

The investigators decided to evaluate the effect of the CC, the most convincing and convenient hormonal treatment, in patients with negative first TESE for NOA. It is of main interest to known if CC could enhance the SRR of a second TESE, that is the ultimate possibility to have their own child for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18-55
* Body Mass Index lower than 35
* Patients with confirmed diagnostic of Non Obstructive Azoospermia based on
* 2 negative spermogram with centrifugation (three month in between)
* Failure of detecting spermatozoid at first testicular sperm extraction (TESE)
* Patients without sperm cells at semen analysis
* Signed informed consent
* Patients benefiting from a social insurance system or a similar system

Exclusion Criteria:

* Patients with grade 2 or 3 varicocele, persistant after cure of the varicocele.
* Patients with current or history of testicular tumor detected on a less than 3 months' ultrasound.
* Patients with history of any other cancer of less than 5 years.
* Patient with Klinefelter or karyotype abnormalities
* Yq micro-deletions
* First TESE conducted under hormonal treatment (Clomifene, Tamoxifen, gonadotrophins or anti-aromatase)
* Patients receiving a treatment known to alter male fertility (see RCP of the treatment, colchicine, methotrexate, ….) in the 6 months before inclusion.
* Patients receiving treatment know to modify the gonadotroph axis activity (FSH, TESTO, DHT, HCG…)
* Hypogonadotropic Hypogonadism
* Persistant bilateral abdominal cryptorchidism
* Patient unable to understand the purpose of the trial or refusing to follow treatment and post-treatment instructions
* Patients with history of psychiatric disorder
* Participation to another trial that would interfere with this trial
* Patients under legal protection

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
presence of sperm cells point of view | 9 months
  Evaluate, versus placebo, the interest of 9 months treatment by 50 mg of Clomiphene citrate to increase the proportion of patient for which at least one sperm cell can be isolated either from the semen at 9 months of treatment or, in case of persistent azoospermia, from a second TESE attempt performed at 9 months of treatment

SECONDARY OUTCOMES:
number of sperm cells point of view | 9 months
  Evaluate, versus placebo, the interest of 9 months treatment by 50 mg of Clomiphene citrate to increase the number of spermatozoa obtained, from the semen at 9 months of treatment or, in case of persistent azoospermia, from a second TESE attempt performed at 9 months of treatment
Follicle Stimulating Hormone (FSH) level evolution | 9 months
  Evaluate the evolution of FSH in both groups
testosterone level evolution | 9 months
  Evaluate the evolution of testosterone in both groups
Luteinizing hormone (LH) level evolution | 9 months
  Evaluate the evolution of LH in both groups
Sex Hormone-Binding Globulin (SHBG) level evolution | 9 months
  Evaluate the evolution of SHBG in both groups
Bioavailable testosterone Inhibin B level evolution | 9 months
  Evaluate the evolution of bioavailable testosterone Inhibin B in both groups
number spermatogonia | 9 months
  Evaluate Hypospermatogenesis status
number of spermatocytes, | 9 months
  Evaluate Hypospermatogenesis status
number of round elongated spermatids | 9 months
  Evaluate Hypospermatogenesis status
prevalence of Sertoli cell only syndrome | 9 months
  Evaluate Sertoli cell only syndrome status
prevalence of maturation arrest | 9 months
  Evaluate maturation arrest status
number of Clomiphene citrate capsules | 9 months
  Compliance will be measured by counting the number of Clomiphene citrate capsules remaining in the brought back at each visit
number of adverse events | 9 months
  Evolution of Clomiphene citrate proportion of side effects
proportion of complications at the second TESE | 9 months
proportion of Pregnancies | 9 months
  proportion of pregnancies after Intracytoplasmic sperm injection
proportion of Miscarriages | 9 months
  proportion of Miscarriages after ICSI
number of Newborn | 9 months
  proportion of Newborn after ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Plotton Ingrid, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Hôpital Femme-Mère-Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No